CLINICAL TRIAL: NCT05223751
Title: Parasympathetic Augmentation Via Respiratory Training for Patients With Systolic Heart Failure
Acronym: PART-HF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment goal was not reached within the allotted funding period.
Sponsor: Lancaster General Hospital (Other)
Collaborators: Louise von Hess Medical Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-XXXX-LGHP
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Diastolic Heart Failure
Keywords: heart failure
MeSH Terms: conditions — Heart Failure, Diastolic; Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRV4 + Breathing and Humming Training (Experimental): On a biweekly basis, and with the other members of their subgroup within the cohort, participants will meet with the Meo Health breathing coach on Zoom for approximately 30 minutes. These sessions will encourage participants to complete their daily exercises and provide additional respiratory training.
  Interventions: Behavioral: Meo Health Breathing and humming exercises
- HRV4 Only (No Intervention): Control participants will complete the daily heart rate variability (HRV) reading using the HRV4Training application.

INTERVENTIONS:
Behavioral: Meo Health Breathing and humming exercises — The Intervention Group will receive training on the Meo Health breathing therapy, which will include:
  * Being shown the Meo Health Breathing Therapy On-Boarding video
  * Orientation to breathing application: Participants will be assisted in downloading and customizing the Breathe application.
  * Zoom tutorial: Participants will be assisted in setting up and navigating Zoom application for use with the Meo Health breathing coach.
  Within one month of the baseline visit, participants in the intervention group will have a 20 minute one-on-one training session with the Meo Health breathing coach. This will mark the beginning of their respiratory training intervention.
  A 3 month visit will occur 3 months (± 14 days) from the one-on-one training session for participants in the intervention group.
  A 6 month visit will occur 6 months (± 14 days) from the one-on-one training session for participants in the intervention group.
  Arms: HRV4 + Breathing and Humming Training

SUMMARY:
This is a prospective, randomized, controlled clinical trial in which participants with NYHA class II or III and symptomatic Heart Failure with reduced Ejection Fraction (HFrEF) (Ejection Fraction (EF) ≤ 45%) will be assigned to one of two treatment groups: standard of care or breathing therapy.

DETAILED DESCRIPTION:
To evaluate the effect of breathing training on the 6-minute walk test in a population of heart failure patients.

Enrollment/Baseline Visit During the enrollment visit, the participant will meet with the clinical research coordinator (CRC) to review any final questions regarding the study and the informed consent form will be signed. The enrollment visit must occur within one month of screening. Once the informed consent is signed, the following procedures will occur.

* Randomization: Participants will be randomized using REDCap in a 2:1 blocking method into the intervention group (breathing therapy) or the control (standard of care).
* N-terminal (NT)-pro hormone BNP (NT-proBNP): If an NT-proBNP was collected as standard of care within 3 months of enrollment, this can be used for study purposes and compared to the 6 month NT-proBNP.
* New York Heart Association Class: If the NYHA class is completed as standard of care within 3 months of enrollment, this can be used for study proposes.
* Kansas City Cardiomyopathy Questionnaire (KCCQ)
* Respiratory Rate
* Peak Expiratory Flow
* 6-minute walk test
* Orientation to the Heart Rate Variability 4 (HRV4) Training application: This will include downloading, creating an account for, and training the participant on the application.

The Intervention Group will also receiving training on the Meo Health breathing therapy, which will include:

* Being shown the Meo Health Breathing Therapy On-Boarding video
* Orientation to breathing application: Participants will be assisted in downloading and custom setting the Breathe application.
* Zoom Within one month of the baseline visit, participants in the intervention group will have a one-on-one training session with the Meo Health breathing coach. This will mark the beginning of their breathing therapy intervention.

  3 Month Visit The 3 month visit will occur 3 months (± 14 days) from the one-on-one training session for participants in the intervention group . The participant will only meet with the CRC at the 3 month visit and all assessments will be completed by the CRC.
* NYHA class
* KCCQ
* Respiratory Rate
* Peak Expiratory Flow
* 6-minute walk test
* Assess compliance from HRV4 Training application questions
* Assess any possible adverse events

  6 Month/Final Visit The 6 month visit will occur 6 months (± 14 days) from the one-on-one training session for participants in the intervention group. The participant will meet with the CRC at the 6 month visit, any assessments not completed as Standard of Care (SOC), will be completed by the CRC.
* NT-proBNP: If an NT-proBNP is ordered as standard of care for the participant, this can be used for study purposes and compared to the baseline NT-proBNP.
* NYHA class: If the NYHA class is completed as standard of care, this can be used for study purposes and compared to the baseline and 3 month values.
* KCCQ
* Respiratory Rate
* Peak Expiratory Flow
* 6-minute walk test
* Assess any possible adverse events

  9 Month Structured Telephone Survey The 9 month structured telephone interview will take place for all participants who receive breathing training from Meo Health. Participants will be called by a study team member who will facilitate a short (3-5 minute) telephone survey about adherence and changes in health outcomes as a result of participation in the trial. (See appendix 15.4). The study team member will record all answers into REDCap. Upon completion of the survey, participants will be closed out of the study. If a study team member is unable to get in contact with a participant after two attempts, their status will be marked as "closed to follow-up" and they won't be interviewed.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Signed informed consent
3. NYHA class II-III heart failure
4. EF ≤ 45% (echo within 1 year of enrollment)
5. At least 30 days of stable medical regimen (no new neurohormonal blockade or Sodium-glucose co-transporter 2 inhibitors (SGLT2i). Dose adjustments allowed)
6. Likely to be compliant with breath training as assessed by the provider
7. Availability of a "smart" phone and internet access
8. Established care at Lancaster General Health Penn Medicine

Exclusion Criteria:

1. Cardiac resynchronization therapy (CRT) within 6 months
2. Severe Chronic obstructive pulmonary disease (COPD)
3. History of diaphragm paralysis
4. Unable or unwilling to complete respiratory training protocol
5. Decompensated or American College of Cardiology (ACC) Stage D Heart Failure (HF)
6. Prior or planned chest/abdominal or nasal/facial surgery within 6 months
7. Neuromuscular disease which impairs respiration
8. Diagnosed cognitive impairment (unable to participate in training)
9. Untreated obstructive severe sleep apnea (AHI > 30)
10. Severe valvular heart disease
11. Uncontrolled atrial fibrillation (Ave Heart Rate (HR) > 100 bpm)
12. Orthopedic or other limitations which impair the 6-minute walk test

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline to 6 months for the 6-minute walk test (6MWT) | Baseline, 6 months
  Distance (m) covered in six minutes from baseline to 6 months

SECONDARY OUTCOMES:
Kansas City Cardiomyopathy Questionnaire 12 (KCCQ12) quality of life score | Baseline, 3 months, 6 months
  Change in Kansas City Cardiomyopathy Questionnaire 12 - Quality of Life (KCCQ12-QL) score
  KCCQ12-QL score corresponds to Questions 6 and 7. Responses are coded as follows:
  Question 6 Response It has extremely limited my enjoyment of life = 1 It has limited my enjoyment of life quite a bit = 2 It has moderately limited my enjoyment of life = 3 It has slightly limited my enjoyment of life = 4 It has not limited my enjoyment of life at all = 5
  Question 7 Response Not at all satisfied = 1 Mostly dissatisfied = 2 Somewhat satisfied = 3 Mostly satisfied = 4 Completely satisfied = 5
  If responses to both questions are missing, no score is computed. Otherwise, the score is calculated by taking the average of the non-missing responses and rescaling to 0-100, as follows:
  KCCQ12-QL = 100*[(average of Questions 6 and 7) - 1]/4
  Scores are scaled 0-100, where 0 denotes the lowest reportable health status and 100 the highest.
Pulmonary parameters: Peak expiratory flow | Baseline, 3 months, 6 months
  Change in peak expiratory flow spirometry
New York Heart Association (NYHA) Class (graded I-IV) Proportion Improved 1 Class | Baseline, 6 months
  Proportion of subjects that decreased 1 NYHA class.
  NYHA Classification - The Stages of Heart Failure:
  Class I - Cardiac disease, but no symptoms and no limitation in ordinary physical activity.
  Class II - Mild symptoms and slight limitation during ordinary activity. Class III - Significant limitation in activity due to symptoms. Comfortable only at rest.
  Class IV - Severe limitations. Symptoms even while at rest. No NYHA class listed or unable to determine.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Small, MD, Principal Investigator — Medical Director
Locations (1):
- Lancaster General Hospital, Lancaster, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No